CLINICAL TRIAL: NCT06212739
Title: Comparison of Post-operative Pain Between Fistula Laser Closure and Ligation of the Intersphincteric Tract in the Treatment of Anal Fistula - a Randomized Controlled Trial. (LASERLIFT)
Brief Title: Post-op Pain After Fistula Laser Closure or Ligation of the Intersphincteric Tract for Anal Fistula
Acronym: LASERLIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MREC 201892-6637
Record Dates: First submitted 2023-12-25; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-12

CONDITIONS: Fistula in Ano
MeSH Terms: conditions — Rectal Fistula | interventions — Lasers

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor was blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser (Experimental): Patients treated using fistula laser closure.
  Interventions: Procedure: Laser
- LIFT (Active Comparator): Patients treated using ligation of intersphincteric fistula tract.
  Interventions: Procedure: LIFT

INTERVENTIONS:
Procedure: Laser — Diode laser used to effect closure of the anal fistula tract
  Other Names: FiLAC
  Arms: Laser
Procedure: LIFT — The intersphincteric portion of the fistula is excised and ligated.
  Other Names: Ligation of the Intersphincteric Fistula Tract
  Arms: LIFT

SUMMARY:
This is a prospective, double-blinded randomised controlled trial conducted at two tertiary hospitals by a credentialed colorectal surgeon.

DETAILED DESCRIPTION:
Patients with high transphincteric fistulas were blinded and randomized to either laser or ligation of the fistula tract (LIFT). Pain scores at rest and movement, at 6 and 24 hours post operatively were measured using the visual analogue scale (VAS). Operative time was measured in minutes Continence and quality of life was assessed via the Wexner incontinence scale and SF-36 questionnaire respectively at 0, 3 and 6 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Complex transphincteric fistulas:
* high transphincteric fistula, involving more than 30% of the external anal sphincter
* Multiple fistulas
* Anterior fistulas
* 18-75 years old
* Able to give consent
* New or recurrent fistulas
* Fistulas with or without setons

Exclusion Criteria:

* Active perianal sepsis requiring drainage
* Fistulas of non-cryptogladular origin- Crohn's, TB, malignancy
* Expected lifespan less than 6 months
* Pregnant women
* Patients with more than 1 definitive surgery done for the fistula before
* Patients with human immunodeficiency virus infection
* Patients with pre-existing chronic pain disorders
* Patients with Non-steroidal Anti-inflammatory Drug (NSAIDS) / Paracetamol allergies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Post-operative pain score | 6 hours, 24 hours
  Post-operative pain will be assessed by a blinded assessor using the Visual Analogue Scale (VAS), a validated pain score.

SECONDARY OUTCOMES:
Operative time | Intraoperative
  Median operative time was to compare the two arms
Continence | At baseline, and at 1 week, 1 month and 6 months post-operatively
  The Wexner score was used to assess pre- and post-operative continence. Minimum score is 3, maximum score is 12. The lower the score, the worse the incontinence.
SF36 | At baseline, and at 1 week, 1 month and 6 months post-operatively
  The SF36 was used to assess pre- and post-operative quality of life.
Return to work | Number of days taken to return to work, assessed at 6 months post-operatively
  Days until return to work
Duration of analgesia use | Number of days until cessation of analgesia use, assessed at 1 week or 1 month, whichever is shorter
  The duration in days that the patient needed to use analgesia post-operative
Failure rate | 6 months
  Failure to heal was defined as failure of fistula closure (persistent discharge) beyond 6 months' post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: April C Roslani, MS, FACS, Principal Investigator — Universiti Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

REFERENCES:
- [Derived] Low JQL, Rajandram R, Aziz MRA, Roslani AC. Postoperative pain following laser fistula closure versus ligation of the intersphincteric fistula tract: A prospective double-blinded randomized controlled trial. World J Surg. 2024 Aug;48(8):1990-1999. doi: 10.1002/wjs.12242. Epub 2024 Jun 6. PMID 38844401

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT06212739/Prot_SAP_000.pdf